The effect of different altitude levels on spinal anesthesia in cesarean section surgery; Comparison of anesthesia parameters and hemodynamic changes

## **INFORMED CONSENT FORM**

This study you participated in is a scientific research and the name of the research is "The effect of different altitude levels on spinal anesthesia in cesarean section surgery; Comparison of anesthesia parameters and hemodynamic changes". The aim of this study is to determine the differences, if any, in terms of anesthetic parameters among pregnant women who underwent cesarean section under neuraxial anesthesia under elective conditions living at different altitudes. The duration of your participation in this research is 1 week.

It is your responsibility to answer only the questions asked in the questionnaire regarding this research. There were no harmful effects for you in this study.

You or your legal representative will be notified immediately of any developments that may be of interest to you during the investigation. For additional information about the research or for any problems, undesirable effects or other discomforts related to the study, Dr.Dilek YENİAY for Giresun University Gynecology and Child Education and Research Hospital, Dr.Selçuk KAYIR for Hitit University Faculty of Medicine. a, You can apply to Dr.Sait Sadi AYDIN for Van Regional Training and Research Hospital.

No payment will be made to you for your participation in this research, and no fee will be charged from you or the social security institution you are affiliated with for all examinations, tests, tests and medical care services within the scope of this research. This research is supported by Giresun University Training and Research Hospital, Hitit University Faculty of Medicine, Van Regional Training and Research Hospital.

Participation in this research is entirely at your own discretion. You can refuse to participate in the research or leave the research at any stage; this will not result in any penalties or impediments to your benefits. The researcher, within your knowledge or against your will, if you do not fulfill the requirements of the treatment scheme, disrupt the work program or increase the effectiveness of the treatment, etc. reasons may exclude you from the study. As stated in Article 22 of Chapter VII of the Biomedicine Convention, "When any part of the human body is removed during an intervention, that part may be stored and used for any purpose other than the purpose for which it was removed only if appropriate information and consent procedures are followed". The results of the research will be used for scientific purposes; In the event that you withdraw from the study or are removed by the investigator, the medical data about you can also be used for scientific purposes, if necessary.

All your medical and identity information will be kept confidential, and your identity information will not be disclosed even if the research is published, but research audiences, pollsters, ethics committees and official authorities can access your medical information when necessary. You can also access your own medical information whenever you want (in case the treatment is confidential, the volunteer should be informed that he/she can access his/her medical information only after the analysis of the data).

## **Consent to Participate in the Study:**

I have read and verbally listened to the above information that should be given to the volunteer before starting the research. I asked all the questions that came to my mind to the researcher, and I understood in detail all the written and verbal explanations made to me. I was given sufficient time to decide whether I wanted to participate in the study. Under these circumstances, I authorize the researcher to review, transfer and process my medical information, and I voluntarily accept the invitation to participate in the research in question without any coercion or pressure.

A signed copy of this form will be given to me.

| Your volunteer | The researcher who made the explanations, |
|---|---|
| Name and surname: | Name and surname: |
| Address: | Mission: |
| TelFax: | Address: |
| | TelFax: |
| Date and Signature: | |
| | Date and Signature: |
| For those under custody or guardianship, the parent or | Institution officer/interview witness who witnessed the consent |
| guardian, | process from the beginning to the end, |
| | Name and surname: |
| Name and surname: | Mission: |
| Address: | Address: |
| TelFax: | TelFax: |